CLINICAL TRIAL: NCT06385106
Title: Effects of Repetitive Transcranial Magnetic Stimulation on Sleep and Cognitive Function in Patients With Alzheimer's Disease: a Randomized, Double-blind, Controlled Study
Brief Title: Effects of Repetitive Transcranial Magnetic Stimulation in Patients With Alzheimer's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: rTMS in AD
Record Dates: First submitted 2024-04-08; First posted 2024-04-25 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease; sleep; Glymphatic System; Transcranial Magnetic Stimulation; cognitive impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Repetitive transcranial magnetic stimulation (Experimental): participants will receive10 sessions of high frequency rTMS treatment applied to the dorsolateral prefrontal cortex over a 5 days real rTMS
  Interventions: Device: Real repetitive transcranial magnetic stimulation
- Sham repetitive transcranial magnetic stimulation (Sham Comparator): participants will receive10 sessions of high frequency rTMS treatment applied to the dorsolateral prefrontal cortex over a 5 days sham rTMS
  Interventions: Device: Sham repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Real repetitive transcranial magnetic stimulation — The target brain region for stimulation was the left dorsolateral prefrontal lobe. The intensity of the stimulation was 80% of the resting motor threshold (MT) of each subject. In the target brain region, we applied 40 stimuli at a frequency of 20 Hz and the MT for 1600 pulses per session.
  Arms: Repetitive transcranial magnetic stimulation
Device: Sham repetitive transcranial magnetic stimulation — The target brain region for stimulation was the left dorsolateral prefrontal lobe. The intensity of the stimulation was 80% of the resting motor threshold (MT) of each subject. In the target brain region, we applied 40 stimuli at a frequency of 20 Hz and the MT for 1600 pulses per session. The patients were applied with the coil angled away from the head to reproduce the noise of the stimulation as well as some local sensation
  Arms: Sham repetitive transcranial magnetic stimulation

SUMMARY:
Previous studies have shown that repetitive transcranial magnetic stimulation (rTMS) can improve cognitive function in Alzheimer's disease (AD), but studies on the improvement of sleep disorders in AD are limited. The aim of this study was to evaluate the effects of rTMS on sleep and cognition in patients with mild-to-moderate Alzheimer's disease (AD).

DETAILED DESCRIPTION:
Transcranial magnetic stimulation (TMS) is a non-invasive brain stimulation technique. Some studies have showed that its positive effects in patients with Alzheimer's disease. The aim of this study was to evaluate the effect of rTMS on sleep and cognitive function in patients with mild to moderate AD, and to evaluate the glymphatic system function's mediating role between sleep and cognitive function. The study involves participants receiving 10 sessions of high frequency rTMS treatment applied to the dorsolateral prefrontal cortex over a 5 days period or sham rTMS. Neuropsychological testing and polysomnography will be used as the primary outcome measures. In addition, magnetic resonance imaging will be used to explore the effect of rTMS on the glymphatic system function in patients with Alzheimer's disease. Follow-up assessments of the patients' status will be conducted at one and three-month intervals.

ELIGIBILITY:
Inclusion Criteria:

1. Participant meets 2014 IWG-2 criteria for hippocampal amnestic syndrome, typical of AD, with progressive episodic memory impairment confirmed by neuropsychology. Cerebrospinal fluid markers (Aβ40, Aβ42, T-tau, p-tau) consistent with AD, or AV-45 PET imaging showing significant cortical tracer retention, in line with AD pathophysiology.
2. Age range: 55-80 years.
3. No visual or hearing impairment.
4. Right-handed.
5. Han nationality.
6. Signed informed consent.
7. Reliable caregivers as information providers.
8. MMSE score: 10-27; CDR: 0.5-2 points.
9. If receiving approved AD treatment (e.g., acetylcholinesterase inhibitor or memantine), dose must be stable for ≥3 months prior to screening and unchanged unless medically necessary.

Exclusion Criteria:

1. History of seizures or epilepsy diagnosis;
2. Stroke history;
3. Nervous system diseases causing brain dysfunction (schizophrenia, severe anxiety/depression, dementia, Huntington's, brain tumors, Parkinson's, metabolic encephalopathy, encephalitis, MS, epilepsy, brain trauma, hydrocephalus);
4. Severe liver/kidney/lung dysfunction, anemia, gastrointestinal disease, arrhythmia, recent MI;
5. Barbiturate/benzodiazepine use within 2 weeks;
6. MRI/TMS contraindications (metallic implants);
7. Systemic diseases causing cognitive impairment (hypothyroidism, folate/B12 deficiency, infections, alcohol/drug abuse);
8. Aphasia, consciousness disturbance, inability to cooperate;
9. TMS/tDCS/DBS has been processed;
10. Underlying pathology other than AD;
11. Focal brain lesions on T1/T2 images;
12. Refusal to sign informed consent.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive funtion | at baseline (T0), immediately after the end of the treatment (T1), 1month later (T2),3months later
  Multidimensional neuropsychological assessment is mainly used to assess the cognitive function of patients. Global cognitive assessment included mini-mental state examination (MMSE) and Montreal Cognitive assessment scale (MoCA). MMSE is widely used in cognitive dysfunction which consists of the following ten parts: orientation, memory, attention and numeracy, ability to recall, language skills, including naming ability, retelling ability, three-step command, reading ability, writing ability. The values range from 0 to 30, with higher score indicating better outcome. MoCA is also an assessment tool for rapid screening of cognitive dysfunction, including 8 cognitive domains such as visual structure skills, executive function, memory, language, attention and concentration, calculation, abstract thinking and orientation. The values range from 0 to 30, with higher score indicating better outcome.
Sleep parameters | at baseline (T0), immediately after the end of the treatment (T1), 1month later (T2),3months later
  Changes in in sleep/wake architecture assessed by polysomnography. Electrodes attached to the scalp near the frontal, central (top) and occipital (back) portions of the brain and provide a readout of different stages of sleep (N1, N2, N3, REM, and Wakefulness). Total sleep time (TST), sleep efficiency (SE), the percentage of rapid eye movement (REM) sleep time in total sleep time, and the percentage of non-rapid eye movement sleep time in total sleep time were mainly analyzed.

SECONDARY OUTCOMES:
glymphatic system | at baseline (T0), immediately after the end of the treatment (T1), 1month later (T2),3months later
  ALPS-index is a non-invasive diffusion tensor image-based method to measure diffusivity along the perivascular space (ALPS), which measures diffusivity in the direction of the perivascular space in the periventricular white matter. It has been proposed to be an indirect indicator of the state of glymphatic function. ALPS-index = mean(Dxxproj; Dxxasso)/mean(Dyyproj; Dzzasso) Dxxproj means diffusivity along the x-axis in the projection fiber. Dxxassoci means diffusivity along the x-axis in the association fiber. Dyyproj means diffusivity along the y-axis in the projection fiber, Dzzassoci means diffusivity along the z-axis in the association fiber. The values was greater than 0 with lower score indicating more damaged.

CONTACTS AND LOCATIONS:
Overall Officials: Benyan Luo, PhD, Study Chair — Zhejiang University
Locations (1):
- The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] You S, Lv T, Qin R, Hu Z, Ke Z, Yao W, Zhao H, Bai F. Neuro-Navigated rTMS Improves Sleep and Cognitive Impairment via Regulating Sleep-Related Networks' Spontaneous Activity in AD Spectrum Patients. Clin Interv Aging. 2023 Aug 15;18:1333-1349. doi: 10.2147/CIA.S416992. eCollection 2023. PMID 37601952
- [Background] Siow TY, Toh CH, Hsu JL, Liu GH, Lee SH, Chen NH, Fu CJ, Castillo M, Fang JT. Association of Sleep, Neuropsychological Performance, and Gray Matter Volume With Glymphatic Function in Community-Dwelling Older Adults. Neurology. 2022 Feb 22;98(8):e829-e838. doi: 10.1212/WNL.0000000000013215. Epub 2021 Dec 14. PMID 34906982
- [Background] Herring WJ, Ceesay P, Snyder E, Bliwise D, Budd K, Hutzelmann J, Stevens J, Lines C, Michelson D. Polysomnographic assessment of suvorexant in patients with probable Alzheimer's disease dementia and insomnia: a randomized trial. Alzheimers Dement. 2020 Mar;16(3):541-551. doi: 10.1002/alz.12035. Epub 2020 Jan 15. PMID 31944580